CLINICAL TRIAL: NCT01910181
Title: A Phase I Open-Label, Multicenter, Multiple-Dose Study to Investigate the Pharmacokinetics, Safety, and Efficacy of Vemurafenib in Chinese Patients With BRAF V600 Mutation-Positive Unresectable or Metastatic Melanoma
Brief Title: A Study of Vemurafenib (Zelboraf) in Chinese Participants With BRAF V600 Mutation-Positive Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO28390
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

ARMS (2):
- Vemurafenib: Pharmacokinetic Cohort (Experimental): Participants will receive vemurafenib orally as 960 mg twice daily on Days 1 to 21 (morning dose only on Day 21), with a drug holiday from Days 22 to 27, and from Day 28 until progression, unacceptable toxicity, consent withdrawal, decision by the investigator or Sponsor, or protocol/eligibility violation.
  Interventions: Drug: Vemurafenib
- Vemurafenib: Expansion Cohort (Experimental): Participants will receive vemurafenib orally as 960 mg twice daily from Day 1 until progression, unacceptable toxicity, consent withdrawal, decision by the investigator or Sponsor, or protocol/eligibility violation.
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Participants will receive vemurafenib at a dose of 960 mg twice daily orally.
  Other Names: Zelboraf

SUMMARY:
This open-label, multicenter study will evaluate the pharmacokinetics, safety and efficacy of vemurafenib in Chinese participants with BRAF V600 mutation-positive unresectable or metastatic melanoma. Participants will receive vemurafenib 960 milligrams (mg) orally twice daily until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female participants, greater than or equal to (≥) 18 years of age
* Histologically confirmed metastatic melanoma (surgically unresectable Stage IIIC or Stage IV, American Joint Committee on Cancer)
* Treatment-naïve or having received prior systemic treatments for metastatic melanoma
* Positive BRAF V600 mutation result determined by a designated laboratory using the Cobas 4800 BRAF V600 Mutation Test
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Previous allowed chemotherapy, immunotherapy, or radiation therapy must have been completed at least 2 weeks prior to study drug administration, and all associated toxicity must be resolved (to less than or equal to [≤] Grade 1 or baseline)
* Recovery from effects of any major surgery (excluding tumor biopsy at baseline) or significant traumatic injury at least 14 days before the first dose of study treatment
* Adequate hematologic, renal, and liver function as defined by protocol
* Fertile men and women must use an effective method of contraception during treatment and for ≥6 months after completion of treatment as directed by their physician (in accordance with local requirements).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than (>) 3 months
* Able to swallow pills

Exclusion Criteria:

* Active central nervous system (CNS) lesions (radiographically unstable/symptomatic lesions), except participants treated with stereotactic therapy or surgery who remain without evidence of disease progression in brain for ≥3 months and have been off corticosteroid and anticonvulsant therapy for ≥3 weeks
* History of or known spinal cord compression or carcinomatous meningitis
* Anticipated or ongoing administration of anti-cancer therapies other than those administered in this study
* Active squamous cell carcinoma (SCC) that has not been excised or has not yet adequately healed post excision
* Pregnant or lactating women
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant small bowel resection that would preclude adequate vemurafenib absorption
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, serious cardiac arrhythmia requiring medication, uncontrolled hypertension, cerebrovascular accident or transient ischemic attack, or symptomatic pulmonary embolism
* Known clinically significant active infection
* History of allogeneic bone marrow transplantation or organ transplantation
* Previous malignancy within the past 5 years other than adequately treated basal cell carcinoma or SCC of the skin, melanoma in-situ, and carcinoma in-situ of the cervix and/or curatively treated cancer from which the participant is currently disease-free, or any malignancy from which the participant has been continuously disease-free for at least 5 years
* Previous treatment with a BRAF inhibitor (sorafenib allowed) or MEK inhibitor
* Participants who have had one or more doses of vemurafenib in a previous clinical trial
* Known human immunodeficiency virus (HIV) positivity or acquired immune deficiency syndrome (AIDS)-related illness, or hepatitis B virus or hepatitis C virus (HCV) carriers (hepatitis B surface antigen-positive, HCV antibody-positive)
* Received any investigational treatment within 4 weeks of study drug start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-08-17 (Actual); Primary Completion 2013-10-22 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing
  - Sun Yet-sen University Cancer Center, Guangzhou

REFERENCES:
- [Derived] Si L, Zhang X, Xu Z, Jiang Q, Bu L, Wang X, Mao L, Zhang W, Richie N, Guo J. Vemurafenib in Chinese patients with BRAFV600 mutation-positive unresectable or metastatic melanoma: an open-label, multicenter phase I study. BMC Cancer. 2018 May 3;18(1):520. doi: 10.1186/s12885-018-4336-3. PMID 29724167

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib: All Participants: Participants were entered into the study into one of two cohorts. Vemurafenib was administered orally as 960 milligrams (mg) twice daily until progression, unacceptable toxicity, consent withdrawal, decision by the investigator or Sponsor, or protocol/eligibility violation. The Pharmacokinetic (PK) Cohort received treatment on Days 1 to 21 (morning dose only on Day 21), with a drug holiday from Days 22 to 27, and resumed treatment on Day 28. The Expansion Cohort received the same regimen from Day 1 onward, without a drug holiday.
Period: Overall Study
Arm/Group | Vemurafenib: All Participants
Started | 46
PK Cohort | 20
Expansion Cohort | 26
Completed | 0
Not Completed | 46
Not completed — Death | 37
Not completed — Lost to Follow-up | 3
Not completed — Study Terminated by Sponsor | 6

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of study medication.
Groups:
- Vemurafenib: All Participants: Participants were entered into the study into one of two cohorts. Vemurafenib was administered orally as 960 mg twice daily until progression, unacceptable toxicity, consent withdrawal, decision by the investigator or Sponsor, or protocol/eligibility violation. The PK Cohort received treatment on Days 1 to 21 (morning dose only on Day 21), with a drug holiday from Days 22 to 27, and resumed treatment on Day 28. The Expansion Cohort received the same regimen from Day 1 onward, without a drug holiday.
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of RO5185426 From 0 to 8 Hours on Day 1
Description: Plasma PK samples were obtained from each participant for calculation of AUC from 0 to 8 hours, using the linear trapezoid rule. The value was averaged among all participants and expressed in hours by micrograms per milliliter (h*μg/mL).
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8 hours) on Day 1
Population: PK Population: All participants who provided evaluable data for PK analysis and did not have a significant protocol violation/deviation.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Groups:
- Vemurafenib: PK Cohort: The PK Cohort was first to recruit. Vemurafenib was administered orally as 960 mg twice daily on Days 1 to 21 (morning dose only on Day 21), with a drug holiday from Days 22 to 27, and from Day 28 until progression, unacceptable toxicity, consent withdrawal, decision by the investigator or Sponsor, or protocol/eligibility violation.
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 20
h*μg/mL | 37.54 (22.31)

2. Primary Outcome: AUC of RO5185426 From 0 to 8 Hours on Day 21
Description: Plasma PK samples were obtained from each participant for calculation of AUC from 0 to 8 hours, using the linear trapezoid rule. The value was averaged among all participants and expressed in h*μg/mL.
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8 hours) on Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
h*μg/mL | 501.28 (122.99)

3. Primary Outcome: AUC of RO5185426 From 0 to 12 Hours on Day 1
Description: Plasma PK samples were obtained from each participant for calculation of AUC from 0 to 12 hours, using the linear trapezoid rule. The value was averaged among all participants and expressed in h*μg/mL.
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12 hours) on Day 1
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
h*μg/mL | 57.51 (32.61)

4. Primary Outcome: AUC of RO5185426 From 0 to 12 Hours on Day 21
Description: as for outcome 3
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12 hours) on Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
h*μg/mL | 720.31 (185.80)

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of RO5185426 on Day 1
Description: Plasma PK samples were obtained from each participant, and the maximum observed post-dose concentration was recorded. The value was averaged among all participants and expressed in micrograms per milliliter (μg/mL).
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12 hours) on Day 1
Population: PK Population.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 20
μg/mL | 6.93 (3.86)

6. Primary Outcome: Cmax of RO5185426 Following Day 21 Dose
Description: Plasma PK samples were obtained from each participant, and the maximum observed post-dose concentration was recorded. The value was averaged among all participants and expressed in μg/mL.
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12, 24, 28, 72, 76, 168 hours) from Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
μg/mL | 77.55 (17.87)

7. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of RO5185426 on Day 1
Description: Plasma PK samples were obtained from each participant, and the time of maximum post-dose concentration was recorded. The median value was derived from all participants and expressed in hours.
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12 hours) on Day 1
Population: PK Population.
Measure: Median (Full Range); unit: hours
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 20
hours | 4.97 [2.0 to 8.0]

8. Primary Outcome: Tmax of RO5185426 Following Day 21 Dose
Description: as for outcome 7
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12, 24, 28, 72, 76, 168 hours) from Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Median (Full Range); unit: hours
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
hours | 1.00 [0.0 to 5.0]

9. Primary Outcome: AUC From 0 to 168 Hours of RO5185426 Following Day 21 Dose
Description: Plasma PK samples were obtained from each participant for calculation of AUC from 0 to 168 hours, using the linear trapezoid rule. The value was averaged among all participants and expressed in h*μg/mL.
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12, 24, 28, 72, 76, 168 hours) from Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
h*μg/mL | 4328.15 (1844.35)

10. Primary Outcome: Elimination Half-Life (t1/2) of RO5185426 Following Day 21 Dose
Description: Plasma PK samples were obtained from each participant for calculation of t1/2, defined as the time elapsed for plasma concentrations to drop by half. The value was averaged among all participants and expressed in hours.
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12, 24, 28, 72, 76, 168 hours) from Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 18
hours | 35.56 (18.06)

11. Primary Outcome: Trough Plasma Concentration (Ctrough) of RO5185426 on Day 15
Description: Plasma PK samples were obtained from each participant, and the concentration immediately prior to drug administration was recorded. The value was averaged among all participants and expressed in μg/mL.
Time Frame: Pre-dose (0 hours) on Day 15
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
μg/mL | 63.000 (23.327)

12. Primary Outcome: Ctrough of RO5185426 on Day 19
Description: as for outcome 11
Time Frame: Pre-dose (0 hours) on Day 19
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
μg/mL | 65.595 (23.645)

13. Primary Outcome: Ctrough of RO5185426 on Day 21
Description: as for outcome 11
Time Frame: Pre-dose (0 hours) on Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
μg/mL | 72.583 (19.979)

14. Primary Outcome: Accumulation Ratio of RO5185426 AUC From 0 to 8 Hours Between Day 21 and Day 1
Description: Plasma PK samples were obtained from each participant for calculation of AUC from 0 to 8 hours, using the linear trapezoid rule. The AUC on Day 21 was divided by the AUC for Day 1. The resulting value was averaged among all participants and expressed as the accumulation ratio.
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8 hours) on Days 1 and 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: accumulation ratio
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 19
accumulation ratio | 17.9 (14.1)

15. Primary Outcome: Terminal Elimination Rate Constant (Kel) of RO5185426 on Day 21
Description: Plasma PK samples were obtained from each participant and the kel was estimated. The value was averaged among all participants and expressed in inverse hours (h^-1).
Time Frame: Pre-dose (0 hours) and post-dose (1, 2, 4, 5, 8, 12, 24, 28, 72, 76, 168 hours) from Day 21
Population: PK Population; only participants who provided sufficient data for the designated timeframe/visit were included.
Measure: Mean (Standard Deviation); unit: hours^-1
Arm/Group | Vemurafenib: PK Cohort
Number analyzed (Participants) | 18
hours^-1 | 0.02 (0.01)

16. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Tumor response was evaluated using RECIST version 1.1 criteria. CR was defined as disappearance of all target lesions and short-axis reduction of any pathological lymph nodes to less than (<) 10 millimeters (mm). PR was defined as greater than or equal to (≥) 30 percent (%) decrease from Baseline in sum diameter of target lesions. The percentage of participants with a best overall response of CR or PR during the study was reported.
Time Frame: Tumor assessments at Screening, Day 1 of Cycle 3, and every two cycles (cycle length of 28 days) thereafter until disease progression (up to 16 months as of data cutoff 15-Dec-2014)
Population: Safety Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 46
percentage of participants | 52.2 [36.95 to 67.11]

17. Secondary Outcome: Percentage of Participants With Disease Progression or Death Among Participants With a Previous Assessment of CR or PR According to RECIST Version 1.1
Description: Tumor response was evaluated using RECIST version 1.1 criteria. CR was defined as disappearance of all target lesions and short-axis reduction of any pathological lymph nodes to <10 mm. PR was defined as ≥30) decrease from Baseline in sum diameter of target lesions. Disease progression was defined as ≥20% increase on-study in sum diameter of target lesions with absolute increase ≥5 mm, or the appearance of new lesion(s). The percentage of participants who died or progressed after CR or PR was reported.
Time Frame: Tumor assessments at Screening, Day 1 of Cycle 3, and every two cycles (cycle length of 28 days) thereafter until disease progression; survival followed every 3 months until discontinuation from study (up to 16 months as of data cutoff 15-Dec-2014)
Population: Safety Population; only participants with a previous response (assessment of CR or PR) were included.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 24
percentage of participants | 54.2

18. Secondary Outcome: Duration of Response According to RECIST Version 1.1
Description: Tumor response was evaluated using RECIST version 1.1 criteria. CR was defined as disappearance of all target lesions and short-axis reduction of any pathological lymph nodes to <10 mm. PR was defined as ≥30) decrease from Baseline in sum diameter of target lesions. Disease progression was defined as ≥20% increase on-study in sum diameter of target lesions with absolute increase ≥5 mm, or the appearance of new lesion(s). Duration of response was defined as the time from initial response of CR or PR to the first event of disease progression or death. Median time to event was estimated using Kaplan-Meier analysis, and the 95% confidence interval (CI) was estimated using the Brookmeyer-Crowley method.
Time Frame: as for outcome 17
Population: Safety Population; only participants with a previous response (assessment of CR or PR) were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 24
months | 9.13 [7.39 to NA] — The upper limit of 95% CI was not reached due to higher number (more than 40%) of censored observations.

19. Secondary Outcome: Percentage of Participants With Death or Disease Progression According to RECIST Version 1.1
Description: Tumor response was evaluated using RECIST version 1.1 criteria. Disease progression was defined as ≥20% increase on-study in sum diameter of target lesions with absolute increase ≥5 mm, or the appearance of new lesion(s). The percentage of participants with death or disease progression during the study was reported.
Time Frame: as for outcome 17
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 46
percentage of participants | 69.6

20. Secondary Outcome: Progression-Free Survival (PFS)
Description: Tumor response was evaluated using RECIST version 1.1 criteria. Disease progression was defined as ≥20% increase on-study in sum diameter of target lesions with absolute increase ≥5 mm, or the appearance of new lesion(s). PFS was defined as the time from treatment start to the first event of disease progression or death. Median time to event was estimated using Kaplan-Meier analysis, and the 95% CI was estimated using the Brookmeyer-Crowley method.
Time Frame: as for outcome 17
Population: Safety Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 46
months | 8.25 [5.65 to 10.94]

21. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants who died during the study was reported.
Time Frame: Throughout treatment (up to 16 months); survival followed every 3 months until discontinuation from study
Population: Safety Population.
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 46
percentage of participants | 80.4

22. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from treatment start to death from any cause. Median time to event was estimated using Kaplan-Meier analysis, and the 95% CI was estimated using the Brookmeyer-Crowley method.
Time Frame: Throughout treatment (up to 16 months); survival followed every 3 months until discontinuation from study
Population: Safety Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib: All Participants
Number analyzed (Participants) | 46
months | 18.7 [12.2 to 20.6]

ADVERSE EVENTS:
Time Frame: Baseline until up to 28 days of last dose
Description: Safety Population.
Arm/Group | Vemurafenib: All Participants
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib: All Participants (N=46)
Uveitis (Eye disorders) | 1
Chest discomfort (General disorders) | 1
Subarachnoid hemorrhage (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib: All Participants (N=46)
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 33
Gingival bleeding (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 11
Toothache (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 19
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 9
Alanine aminotransferase increased (Investigations) | 7
Amylase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 7
Blood albumin decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 27
Blood bilirubin unconjugated increased (Investigations) | 4
Blood cholesterol increased (Investigations) | 27
Blood lactate dehydrogenase increased (Investigations) | 9
Gamma-glutamyltransferase increased (Investigations) | 12
Low density lipoprotein increased (Investigations) | 8
Protein total decreased (Investigations) | 3
Total bile acids increased (Investigations) | 12
Urobilinogen urine increased (Investigations) | 6
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 34
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 13
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25
Haemoglobinuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 25
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 31
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 5
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5
Palmer-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 19
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13
Skin disorder (Skin and subcutaneous tissue disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Gingival pain (Gastrointestinal disorders) | 4
Gingival ulceration (Gastrointestinal disorders) | 3
Chest discomfort (General disorders) | 4
Gingivitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 6
Blood creatine phosphokinase increased (Investigations) | 3
Blood triglycerides increased (Investigations) | 5
White blood cell count decreased (Investigations) | 3
Protein urine present (Investigations) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT01910181/Prot_SAP_000.pdf